CLINICAL TRIAL: NCT00484081
Title: Prospective Evaluation of Microdissection Testicular Sperm Extraction in Non-Obstructive Azoospermic Men and Their IVF-ICSI Related Outcomes at ART Treatment.
Brief Title: Microdissection Testicular Sperm Extraction (MicroTESE) and IVF-ICSI Outcome in Non-Obstructive Azoospermia (NOA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinic and Research Center in Human Reproduction Roger Abdelmassih (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RA9969
Record Dates: First submitted 2007-06-06; First posted 2007-06-08 (Estimated); Last update posted 2007-06-08 (Estimated); Status verified 2007-06

CONDITIONS: Azoospermia; Infertility
Keywords: TESE; NON-OBSTRUCTIVE; MICRODISSECTION; AZOOSPERMIA; ICSI
MeSH Terms: conditions — Azoospermia; Infertility | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Microdissection Testicular Sperm Extraction
Procedure: ICSI

SUMMARY:
We evaluated the application of surgical testicular exploration with the aid of a microscope (MictoTESE) to increase the chances of obtaining sperm in men with impaired sperm production, a condition known as non-obstructive azoospermia.

We also evaluated the outcomes of these couples when the sperm obtained were used in ICSI (Intracytoplasmic Sperm Injection) during assisted reproductive technology treatment.

We believe that excellent results may be obtained with the use of the following techniques in the treatment of couples where non-obstructive azoospermia is a significant cause.

DETAILED DESCRIPTION:
Men diagnosed with non-obstructive azoospermia and seeking assisted reproductive technology treatment (ART) are candidates for surgical sperm retrieval with the aid of microdissection. We believe that this approach may currently be the best option for these subjects.

We evaluated our surgical sperm retrieval rate associated to their serum LH, FSH, TOTAL TESTOTERONE and PROLACTIN levels, pre-operative testicular volume and also compared to the post-operative histological analysis of fixed testicular tissue specimens collected during the procedure, stained with haematoxylin and eosin.

We also evaluated the outcomes using ICSI based ART for these couples observing mean ICSI and fertilized oocytes, number and quality of embryos transferred, implantation and pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

* Men undergoing ART treatment with clinical diagnosis of non-obstructive azoospermia.
* Female partner undergoing ICSI based ART treatment

Exclusion Criteria:

* Men where non-obstructive azoospermia was not confirmed based on histological analysis of fixed testicular tissue specimens collected by open surgical testicular biopsy and stained with haematoxylin and eosin.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2005-06; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Sperm retrieval rate,mean male and female partner age,mean ICSI and fertilized oocytes, implantation, pregnancy and miscarriage rates.Testicular histology was also compared. | 17 months

SECONDARY OUTCOMES:
Sperm retrieval associated to pre-operative serum FSH, LH, Total Testosterone,Prolactin, testicular volume and post-operative testicular histology. ICSI and pregnancy results associated to sperm motility. | 17 months

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Ravizzini, Dr., Principal Investigator — Clinic and Research Center in Human Reproduction Roger Abdelmassih
Locations (1):
- Clinic and Research Center in Human Reproduction Roger Abdelmassih, São Paulo, São Paulo, Brazil